CLINICAL TRIAL: NCT02469207
Title: A Study Utilising Tissue From Deceased Organ Donors to Investigate Regenerative Cellular Therapies and Related Physiological and Developmental Processes
Brief Title: Regenerative Cellular Therapies, Physiology, Pathology and Developmental Biology
Acronym: RCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Cambridge Stem Cell Institute, Cambridge (Unknown); Anne McLarent Laboratory of Regenerative Medicine, Cambridge (Unknown); The Gurdon Institute, Cambridge (Unknown); Sanger Institure, Cambridge (Unknown); Institute of Metabolic Science, Cambridge (Unknown); MRC Mitochondrial Biology Unit, Cambridge (Unknown)
Responsible Party: Principal Investigator, Dr. Kourosh Saeb-Parsy, Mr Kourosh Saeb-Parsy, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A093532; 15/EE/0152 (Other: Research Ethics Committee)
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Graft Rejection; Transplantation; Diabetes Mellitus
Keywords: regenerative medicine; stem cells; immunomodulatory; induced pluripotent stem cells; gut physiology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA data from tissue samples from donated organs may be retained anonymously for a period up to 10 years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deceased organ donors: Patients with consent for organ donation towards transplantation and research. Organs not used for transplantation will be used for this study if determined appropriate and necessary.
  Interventions: Other: Removal of tissue post-mortem

INTERVENTIONS:
Other: Removal of tissue post-mortem

SUMMARY:
This study aims to use tissue from deceased organ donors to investigate organ physiology, developmental biology, as well as the development of future regenerative cellular therapies. It will investigate function and immune response to stem cells as well as their generation from adult cells and generation of induced pluripotent stem cells (iPSCs).

DETAILED DESCRIPTION:
The purpose of this study is to use tissue from deceased organ donors to address questions that are of importance for the development of regenerative cellular therapies for better understanding of organ physiology and developmental biology. This study aims to maximise the clinically available data as well as patient benefit that can be generated from donated tissue. It also aims to reduce number of consent forms given to patients by consolidating and coordinating a number of related investigations.

The study aims are:

* To examine function and the immune response to stem cells and their differentiated progeny as well as development of immunomodulatory approaches to prevent their rejection.
* Generation of induced pluripotent stem cells (iPSCs) and their subsequent differentiation into functional cells as potential therapies.
* Generation of differentiated cells from native adult stem cells as cellular therapies.
* Investigation of organ physiology.

ELIGIBILITY:
Inclusion Criteria:

* All deceased organ donors with informed consent from the donor family

Exclusion Criteria:

* Donors aged <16

Ages: 16 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All deceased organ donors for whom informed consent is available from the donor family
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of donors from which induced Pluripotent Stem Cells were generated | 5 years

SECONDARY OUTCOMES:
Number of stem cell lines for which the immune response was characterised | 5 years
Number of immunomodulatory therapies characterised | 5 years
Levels of baseline and stimulated gut hormones detected | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Saeb-Parsy, PhD, FRCS, Principal Investigator — Cambridge Univeristy Hospitals
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom